CLINICAL TRIAL: NCT05645575
Title: Pilot Study: Evaluating the Feasibility of Accelerated rTMS Treatment Delivered at Individual Resonant Frequencies for In-patient Subjects Suffering From Major Depressive Disorder
Brief Title: In-patient SCC TMS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Andrew F. Leuchter, Director of the Neuromodulation Division at the Semel Institute, University of California, Los Angeles
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 22-000810
Record Dates: First submitted 2022-12-01; First posted 2022-12-09 (Actual); Last update posted 2025-09-23 (Actual); Status verified 2025-09

CONDITIONS: Major Depressive Disorder
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Intervention Model Description: Open-label Transcranial Magnetic Stimulation Treatment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Open-label TMS (Experimental)
  Interventions: Device: Open-label TMS

INTERVENTIONS:
Device: Open-label TMS — Customized, Open-Label Transcranial Magnetic Stimulation
  Other Names: Transcranial Magnetic Stimulation

SUMMARY:
The investigators are studying the feasibility, safety, and tolerability of administering accelerated repetitive Transcranial magnetic stimulation(a-rTMS) at frequencies other than standard 10 Hz for in-patient Subjects diagnosed with Major Depressive Disorder. Participants will be recruited from the Resnick Neuropsychiatric Hospital. This study will enroll 30 participants who will undergo up to three brain activity recordings, one MRI scan, one TMS procedure to determine the appropriate frequency and intensity for treatment, daily symptom assessments, and 25 TMS treatments. Participants will be asked to participate for up to 2 weeks.

DETAILED DESCRIPTION:
Repetitive Transcranial Magnetic Stimulation (rTMS) is an efficacious treatment for Major Depressive Disorder (MDD) and may hold therapeutic potential for suicidality, specifically. The clinical benefit of rTMS is thought to depend upon successful engagement of brain functional networks, which in turn depends on the preferred oscillatory frequency of the target network for that individual.

The investigators have developed a novel interrogation method to identify the optimal individual stimulation frequency for each participant to enhance treatment response by maximizing the engagement of the functional brain networks. Our data suggest that stimulation at individualized frequencies results in about 50% better response for depression compared to the standard treatment of 10 Hz stimulation. Additionally, an accelerated administration of rTMS (a-rTMS) has been shown safe and tolerable, which is highly desirable in the context of a hospitalization.

The investigators propose to use this approach to administer 25 sessions of individualized a-rTMS left dorsolateral prefrontal cortex (DLPFC) over a course of five days to obtain an accelerated relief of depression symptoms and reduce suicide risk. The investigators will enroll 30 in-patients undergoing treatment in the Resnick Neuropsychiatric Hospital. Patients will first undergo a brief (10-15 min) magnetic resonance imaging (MRI) for the purpose of neuronavigation to the optimal anatomical site. Subsequently, a motor threshold will be identified to determine the optimal stimulation intensity. Patients will receive 5 a-rTMS sessions daily for five days with a minimum interval of 1 hour between sessions. In addition to establishing tolerability and acceptability of the intervention, the goal is to evaluate the preliminary efficacy for improving depressive and suicidality symptoms. The investigators expect the treatment to be well tolerated, providing fast relief of depression and suicidal symptoms.

ELIGIBILITY:
Inclusion Criteria:

1. All subjects must be between 18-65 years of age.
2. Must have confirmed diagnosis of moderate to severe Major Depressive Disorder (single or recurrent episode) as defined by a HAM-D score of 17 or higher.
3. Failure to respond to a minimum of 2 trials of antidepressant medication
4. Failure to respond from at least two different agent classes
5. Accompanied by at least two evidence-based augmentation therapies (Benzodiazepines do not count).
6. Must have a trial of psychotherapy known to be effective in the treatment of MDD of an adequate frequency and duration.
7. Subjects are willing and able to adhere to the accelerated treatment schedule.

   Exclusion Criteria:
8. Are mentally or legally incapacitated, unable to give informed consent
9. Have an infection or poor skin condition over the scalp where the device will be positioned
10. Have increased risk of seizure because of family history, stroke, or currently use medications that lead to increased risk for seizure
11. Diagnosis of acute or chronic psychotic symptoms or disorders (such as schizophrenia, schizophreniform or schizoaffective disorder) in the current depressive episode.
12. Neurological conditions that include epilepsy, cerebrovascular disease, dementia, increased intracranial pressure, having a history of repetitive or severe head trauma, or with primary or secondary tumors in the central nervous system.
13. Presence of an implanted magnetic-sensitive medical device present in the body scan, including but not limited to a cochlear implant, implanted cardioverter defibrillator, pacemaker, vagus nerve stimulator, or metal aneurysm clips or coils, staples, or stents. (Note: Dental amalgam fillings are not affected by the magnetic field and are acceptable for use with transcranial magnetic stimulation and MRI.)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-04-01 (Actual); Primary Completion 2027-02-22 (Estimated); Study Completion 2027-02-22 (Estimated)

PRIMARY OUTCOMES:
Treatment Efficacy as Measured by Change in Inventory of Depressive Symptoms (Self-Report) at Baseline and Final Visit | 2 Weeks (Baseline and Final Visit)
  Treatment efficacy as measured by change in Inventory of Depressive Symptoms (Self-Report) at Baseline and Week 8 visit. This is a 30-item questionnaire with minimum and maximum score values ranging from 0 to 84. Higher scores indicate a worse outcome and lower scores indicate better outcome.

SECONDARY OUTCOMES:
Treatment Efficacy as Measured by Change in Patient Health Questionnaire-9 (PHQ-9) at Baseline and Final Visit. | 2 Weeks (Baseline and Final Visit)
  Treatment efficacy as measured by change in Patient Health Questionnaire-9 (PHQ-9) at Baseline and Final Visit. This is a 9-item questionnaire with minimum and maximum score values ranging from 0 to 27. Higher scores indicate a worse outcome and lower scores indicate better outcome.

CONTACTS AND LOCATIONS:
Locations (1):
- UCLA TMS Service and Research Service, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: Yes
Sharing is dependent on request by other researchers and relation to study condition and treatment. De-identified study data will be shared at the PI's discretion.
Supporting Information: SAP